CLINICAL TRIAL: NCT01654094
Title: A Multicenter, Prospective, Randomized Study to Compare Milliken Dressing P6 to Mafenide Acetate 5% Solution as a Split Thickness Skin Graft Cover Dressing in Burn Wound Patients.
Brief Title: Study of Low Adherent Dressing Versus the Standard of Care for the Management of Skin Grafts Over Thermal Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milliken Healthcare Products, LLC (Industry)
Collaborators: Criterium, Inc. (Industry); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MHP-P6-1; W81XWH-10-2-0159 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2012-07-24; First posted 2012-07-31 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Burns; Skin Burn Requiring Skin Graft
MeSH Terms: conditions — Burns | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- P6 Low Adherent Dressing (Experimental): All participants will serve as their own control. All participants will receive both the P6 Low Adherent Dressings and the Standard of Care (SOC).
  Interventions: Device: P6 Low Adherent Dressing
- Standard of Care (SOC) (Active Comparator): All participants will serve as their own control. All participants will receive both the P6 Low Adherent Dressings and the Standard of Care (SOC).
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Device: P6 Low Adherent Dressing — Each patient will have two similar, non-adjacent study sites. One site will be treated with P6 Low Adherent Dressing and the other site will be treated with the Standard of Care (SOC).
  Arms: P6 Low Adherent Dressing
Other: Standard of Care (SOC) — Each patient will have two similar, non-adjacent study sites. One site will be treated with P6 Low Adherent Dressing and the other site will be treated with the Standard of Care (SOC).
  Arms: Standard of Care (SOC)

SUMMARY:
The purpose of this study is to evaluate the P6 Low Adherent Study Dressing relative to the Standard of Care (SOC, Mafenide Acetate 5% Solution) for the management of skin grafts in burn wounds resulting from thermal burn injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have thermal burns from scalds, flame/fire or contact with a hot object.
* Patients must have a TBSA burn of less than or equal to 50%.
* Patients must have two nonadjacent study burn sites (i.e., separated in such a way that SOC dressing does not contaminate the study dressing) of comparable size (up to approximately 2% TBSA) and severity requiring excision and grafting.
* Patients must have undergone excision and autografting on or before post-burn day (PBD) 14.
* Patients' study burn sites will be treated with skin grafts with a mesh ratio up to 3:1, at the surgeon's discretion.
* Patients expected to be available for assessment of study burn sites at least until POD 6 ±1 day.
* Males or females at least 18 years of age but no older than 65 years of age at the time of informed consent.
* Patient and / or Legally Authorized Representative (LAR) voluntarily agrees to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

* Patients with electrical or chemical burns.
* Patients with a study burn site excised and "grafted" with Integra.
* Patients with study burn sites on the buttocks, scalp, hands, feet, neck or ears.
* Patients taking vasopressors or inotropes.
* Patients using systemic immunosuppressants (e.g., corticosteroids and anti-neoplastic agents, etc.).
* Patients with acute renal failure, defined as creatinine clearance (CrCL) >2.5 mg/dL or AKIN score greater than or equal to 2 or estimated GFR < 30, if the assessment is conducted as part of the patient's routine clinical care.
* Patients with acute respiratory distress syndrome (ARDS), if the assessment is conducted as part of the patient's routine clinical care.
* Patients with liver cirrhosis (Childs-Pugh B Class or greater) or who have AST / ALT levels greater than or equal to 2 times the upper limit of theinstitution's normal range, if the assessment is conducted as part of the patient's routine clinical care.
* Patients with a known sensitivity or known intolerance to mafenide acetate (Sulfamylon) or to silver.
* Patients with any concurrent medical condition, which in the opinion of the investigator, may compromise their safety or the objectives of the study.
* Patients who are breastfeeding, pregnant or expecting to become pregnant during the study..
* Patients who have been exposed to an investigational drug or device within 30 days prior to Screening or is scheduled to receive another investigational drug or device during either the Treatment Phase or Follow-up Evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Management of skin grafts as determined by investigator's visual assessment of percent graft take | 6 days

SECONDARY OUTCOMES:
The incidence of post-operative graft infections | 15 days
Assessment of patient's pain / discomfort, using a visual analog scale. | 15 days
Costs of study burn site wound dressing regimens. | 15 days
Ease of use and clinician preference of the study burn site wound dressing regimens | 15 days
Statistical robustness of visual graft take assessments in-person and from digital photographs | 15 days
Progression of percent graft take with time for both P6 and SOC. | 15 days
Assessment of the incidence and severity of SAEs and wound specific AEs, including local reactions. | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cairns, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - Shands at University of Florida, Gainesville, Florida
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Tennessee Firefighter's Regional Burn Center, Memphis, Tennessee